CLINICAL TRIAL: NCT03886571
Title: U01-Biomarkers for Noninvasive and Early Detection of Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Collaborators: Baylor Research Institute (Other)
Responsible Party: Principal Investigator, Michael Demeure, MD, Program Director for Precision Medicine, Hoag Memorial Hospital Presbyterian
Other Study IDs: 119-17-CA
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Up to 60 mL of blood will be obtained at study entry. Archived paraffin embedded blocks of both normal and tumor tissue and Up to 0.5 mL Pancreatic cyst fluid may be collected if the participant is undergoing an endoscopic or surgical procedure for a pancreatic cyst.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational, biospecimen collection protocol to develop a bank of pancreatic cancer tissue and normal tissue.

DETAILED DESCRIPTION:
This is an observational, biospecimen collection protocol to develop a bank of pancreatic cancer tissue, normal tissue. Biospecimens collected through this protocol will be shared with collaborators in the Pancreatic Cancer Detection Consortium to support projects funded through an NIH U01 grant. Participants will be enrolled when they present for clinically indicated surgical procedures for their possible tumor or pancreas resection or cyst resection, or at a clinically indicated follow-up appointment after their procedure.

This protocol supports this effort by providing investigators with access to a wide variety of pancreatic tissues and biospecimens for translational studies in pancreatic cancer. This protocol covers the collection of clinical data and biospecimens (blood; malignant, benign, or precancerous pancreatic tumor; and adjacent normal tissues) from patients with, or suspected to have, pancreatic cancer. Additionally, saliva and cyst fluid, may be collected in the future from patients with pancreatic cysts. These will be shared with the Pancreatic Cancer Detection Consortium for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females ≥ 18 years of age who have been diagnosed with Pancreatic Cancer (PDAC), Pancreatic Neoplasms (PNs - IPMMs, PanINs and MCNs), pancreatitis and diabetes or no disease/healthy.
* Individuals undergoing or have previously undergone a diagnostic procedure (i.e. EUS or ERCP) evaluation or surgery.
* Willingness and ability to donate biospecimens for the purpose of research.
* Subjects must have had diagnostic procedure or surgery after September 1, 2017.

Exclusion Criteria:

* Individuals under 18 years of age.
* Inability to donate biospecimens.
* Females pregnant or lactating.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with an upcoming standard of care clinical and/or surgical event who meet criteria for study participation are identified by the treating physician and will be asked to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2023-09-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Measuring cell-free and exosomal-miRNA biomarkers using small RNA-Seq in matched tissue and plasma from patients with PDAC, PNs, pancreatitis and normal pancreas for early detection. | 5 years
  We will perform whole genome small RNA sequencing (small RNA-Seq) analysis on tissue specimens from 60 primary PDACs (30 stage I/II and 30 Stage III/IV), 60 PNs (20 each PanINs, IPMNs and MCNs), and 60 non-neoplastic normal pancreatic tissues (NN) and pancreatitis.
  We will perform small RNA-Seq analysis to identify differentially expressed cell-free and exosomal miRNAs (cf-miRNAs and exo-miRNAs) from the same matched plasma specimens.

CONTACTS AND LOCATIONS:
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No